CLINICAL TRIAL: NCT06871280
Title: Assessment of Vertigo and Dizziness in Individuals Following COVID-19
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstanbulPMRTRH222
Record Dates: First submitted 2025-03-10; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study aimed to assess the prevalence of dizziness/vertigo in individuals following COVID-19 and to investigate potential risk factors associated with these symptoms. A total of 296 patients aged 20-66 years who had recovered from COVID-19 were evaluated at Istanbul Physical Medicine and Rehabilitation Training and Research Hospital between June 1, 2021, and December 31, 2021. Clinical and demographic data, including COVID-19 history, comorbidities, and symptom characteristics, were collected. Dizziness-related disability was assessed using the Dizziness Handicap Inventory (DHI), while balance performance was evaluated with the Berg Balance Scale (BBS).

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20-66 years.
* History of confirmed COVID-19 infection.
* Ability to speak and understand Turkish.
* Willingness to provide verbal and written informed consent.

Exclusion Criteria:

* Pre-existing vertigo or balance disorders (e.g., benign paroxysmal positional vertigo, Ménière's disease, vestibular migraine, vestibular neuritis).
* Inner ear diseases or vestibular dysfunction.
* Neurological disorders affecting balance (e.g., multiple sclerosis, Parkinson's disease, history of stroke, epilepsy).
* Psychiatric conditions that could cause dizziness (e.g., anxiety, panic attacks, depression).
* History of head or neck trauma in the past six months.
* Moderate to severe visual impairment.
* Chronic alcohol or substance use.
* Use of ototoxic medications.
* Severe cardiovascular diseases (e.g., orthostatic hypotension, advanced heart failure, severe arrhythmias).
* Pregnant or breastfeeding women.
* Acute infection other than COVID-19 in the past three months.
* Severe COVID-19 requiring hospitalization

Ages: 20 Years to 66 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included 296 patients aged 20-66 years who had recovered from COVID-19 and presented to the outpatient clinic
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | 0 day
  Prevalence of dizziness/vertigo in individuals following COVID-19, assessed using the Dizziness Handicap Inventory (DHI).
  Range: 0-100 (Higher scores indicate greater dizziness-related disability).

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 0 day
  Balance status evaluated using the Berg Balance Scale (BBS). Range: 0-56 (Higher scores indicate better balance)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)